CLINICAL TRIAL: NCT01945437
Title: Magnesium and TKA Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Kim Mihyun, Doctor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Mg_TKA
Record Dates: First submitted 2013-09-13; First posted 2013-09-18 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Control (Placebo Comparator): Control group receive same volume of normal saline as in the magnesium group
- magnesium (Experimental): This group receive magnesium sulfate perioperatively.
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Magnesium Sulfate — The magnesium group receive intravenous magnesium sulfate.
  Arms: magnesium

SUMMARY:
The hypothesis of this study is that in staged bilateral total knee arthroplasty (TKA, magnesium sulfate administered during the perioperative period of the first TKA may decrease pain after the second TKA. It is known that pain is greater in the second TKA than in the first. Therefore, we compared pain of the second TKA between the magnesium and control groups.

ELIGIBILITY:
Inclusion Criteria: American society of anesthesiologist physical status 1 - 2. patients scheduled to undergo staged bilateral TKA

Exclusion Criteria: American society of anesthesiologist physical status >3

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Pain | from the end of the TKA until 48 hour
  Pain measured with visual analogue scale (VAS)

SECONDARY OUTCOMES:
analgesic | from the end of the TKA until 48 hours
  analgesic consumptions from the end of the TKA until 48 hours